CLINICAL TRIAL: NCT02576964
Title: An Open-Label Phase II Study of Capecitabine in Combination With Pegylated Interferon Alfa-2a in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Capecitabine (Xeloda) and Peginterferon Alfa-2a (Pegasys) in Treatment-Naive Participants With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18269
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Capecitabine; peginterferon alfa-2a

ARMS (1):
- Capecitabine + Peginterferon alfa-2a (Experimental): Treatment-naive participants with advanced liver cancer will receive combination treatment with capecitabine (1000 milligrams per meter-squared [mg/m^2] twice daily orally on Days 1 to 14 of each 21-day cycle) and peginterferon alfa-2a (180 micrograms (mcg) subcutaneous [SC] every week during each 21-day cycle) until at least 6 cycles (18 weeks) or disease progression, intolerable toxicity, or consent withdrawal.
  Interventions: Drug: Capecitabine; Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Capecitabine — Participants will receive oral capecitabine, 1000 mg/m^2 twice daily on Days 1 to 14 of each 21-day cycle, for at least 6 cycles (18 weeks). Treatment may continue until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: Xeloda
Drug: Peginterferon alfa-2a — Participants will receive SC peginterferon alfa-2a, 180 mcg every week during each 21-day cycle, for at least 6 cycles (18 weeks). Treatment may continue until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: Pegasys

SUMMARY:
This study will evaluate the efficacy and safety of capecitabine (Xeloda) in combination with peginterferon alfa-2a (Pegasys) in participants with advanced liver cancer who have had no prior treatment. The anticipated time on study treatment is until disease progression, and the target sample size is 43 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 75 years of age
* Locally advanced or metastatic liver cancer with measurable disease and not eligible for any standard therapy

Exclusion Criteria:

* Previous treatment for liver cancer
* Main portal vein involvement
* Bone, brain, or leptomeningeal metastasis
* Clinically significant cardiac disease
* Malabsorption syndrome or lack of physical integrity of the upper gastrointestinal tract
* History of other cancer, except basal cell skin cancer or in situ cancer of the cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | up to post-chemotherapy follow-up ( approximately 46 months)

SECONDARY OUTCOMES:
Time to disease progression | Up to approximately 46 months
Duration of response | Up to approximately 46 months
Overall survival | Up to approximately 46 months
Incidence of adverse events | Up to approximately 46 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- China (2):
  - Beijing
  - Guangzhou
- Taiwan (2):
  - Kueishan
  - Tainan
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla